CLINICAL TRIAL: NCT04234867
Title: A Randomized, Double-Blinded, Placebo-controlled, Single-center Phase 1 Pilot Study to Explore the Effect of DAPAglifozin and Stress ( i.v. ACTH) on the Development of DKA After Insulin Withdrawal in Adolescent and Adult Subjects With T1D
Brief Title: Study to Explore the Effect of Dapagliflozin and Stress in Adolescent and Adult Subjects With Type 1 Diabetes (T1D)
Acronym: Dapa-Stress
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Kinderkrankenhaus auf der Bult (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ESR-17-13152
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes; Diabetic Ketoacidosis
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetic Ketoacidosis | interventions — dapagliflozin; adrenocorticotropin zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dapagliflozin - Stress (Experimental): Administration of 10mg dapagliflozin oral for 5 days and one i.v. administration of 250µg ACTH (Synacthen)
  Interventions: Drug: Dapagliflozin; Other: Stress
- Dapagliflozin and Placebo Stress (Experimental): Administration of 10mg dapagliflozin oral for 5 days and one i.v. administration of Placebo matching Synacthen
  Interventions: Drug: Dapagliflozin; Other: Placebo Stress
- Placebo Dapagliflozin and Stress (Placebo Comparator): Administration of placebo oral for 5 days identical to dapagliflozin and one i.v. administration of 250µg ACTH (Synacthen)
  Interventions: Drug: Placebo oral tablet; Other: Stress
- Placebo Dapagliflozin and Placebo Stress (Placebo Comparator): Administration of placebo oral for 5 days identical to dapagliflozin and one i.v. administration of Placebo matching Synacthen
  Interventions: Drug: Placebo oral tablet; Other: Placebo Stress

INTERVENTIONS:
Drug: Dapagliflozin — once daily for 5 days
  Other Names: Forxiga
  Arms: Dapagliflozin - Stress; Dapagliflozin and Placebo Stress
Drug: Placebo oral tablet — once daily for 5 days
  Other Names: Control
  Arms: Placebo Dapagliflozin and Placebo Stress; Placebo Dapagliflozin and Stress
Other: Stress — single dose after last administration of experimental drug
  Other Names: Synacthen
  Arms: Dapagliflozin - Stress; Placebo Dapagliflozin and Stress
Other: Placebo Stress — single dose after last administration of experimental drug
  Other Names: Stress Control
  Arms: Dapagliflozin and Placebo Stress; Placebo Dapagliflozin and Placebo Stress

SUMMARY:
Type 1 Diabetes is characterized by an absolute lack of insulin caused by autoimmune ß-cell destruction. Looking for different therapeutic approaches, beyond the administration of Insulin SGLT-Inhibitors (SGLT=sodium-glucose cotransporter) like Dapagliflozin look like a promising option to avoid hyperglycaemic excursions which are a reason for glycaemic variability by renal excretion of excessive glucose without administration of extra insulin. But also euglycemic DKA has been reported during SGLT2 add-on therapy to insulin in T1D and mechanistic studies have been called for.

The role of Dapagliflozin-induced hyperglucagonemia and stress/infection precipitating euglycemic DKA in this situation is unclear.

Thus the purpose of this pilot study is to collect clinical data on the development of DKA after insulin-withdrawal with Dapagliflozin compared to placebo and the added effect of a single dose of 4mg/kg i.v. ACTH as mediator of stress.

The first objective is to investigate the time to DKA (defined as Bicarbonate <19 mmol/l) after insulin withdrawal during treatment with a stable 5 day single daily dose of 10mg Dapagliflozin in patients with type 1 Diabetes.

In addition it should be evaluate the additional effect of stress, modelled by a single injection of ACTH on DKA development during Dapagliflozin Treatment.

We also want to know if Dapagliflozin influences glucagon levels during insulin withdrawal and how this is associated with the time course of DKA development.

DETAILED DESCRIPTION:
The purpose of the Dapastress trial is, to evaluate if some metabolic parameters can be identified as an early marker or contributor in development of ketonic metabolic imbalance. As the hormonal "background" is completely different in pubertal adolescents compared to adults (especially contra-insulin hormones as growth hormone, glucagon).

Approximately 20 subjects 18-45 years will be screened in order to randomize 16 patients, where stress and Dapagliflozin (or corresponding placebo) will be administered independently.

The trial will consist of 14 visits: a screening visit (Visit 1), 4 overnight visits complexes (Visit 2 to Visit 13), including phone visits and a follow-up visit (Visit 14). Furthermore, an information visit will take place prior to the screening visit in order to obtain patient's informed consent. Screening will take place 2-21 days prior to Visit 2. The follow-up visit will take place 5-21 days after the end of Visit 13. The overnight visits will be separated by a wash-out period (5-30 days between the end of each visit complex and start of next complex) during which the subjects will resume their normal insulin treatment. Each phone visit will take place 3-5 days after the end of overnight Visits.

The planned total duration of the trial is 58-100 days per subject (rescheduled visits excluded). Each subject will be randomised to a unique treatment sequence (1:1:1:1).

Seq 1: A D B C Seq 2: B A C D Seq 3: C B D A Seq 4: D C A B (e.g. A Dapa-Stress, B Dapa-Placebo Stress , C Placebo- Stress, D Placebo-Placebo Stress)

After randomization patients will receive Dapagliflozin/placebo for 5 single daily Dosis. During the overnight visits the metabolic control will be achieved by a variable i.v. Infusion of human Insulin by an Infusion pump. The procedure will be used in order to aim and maintain blood glucose levels between 70 and 180 mg/dl. The fluid Infusion and Insulin dosing scheme will depend on Body weight and blood glucose levels. At approximately 03:00 hours in the morning the blood glucose should be within target range. Then insulin infusion will be suspended. In the morning the last dose of actual study medication (Dapagliflozin/ Placebo) and the single dose of stress (ACTH or placebo) will be administered. During now started stress phase blood samples for determination of metabolic Panels,blood gas analysis, Glucose and ketone will be taken hourly and vital signs tested. 12 hours after administration of stress (ACTH or placebo) the patients will resume their CSII and will be discharged when being well on investigator's judgement.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent from participant and all legal representatives prior to any study specific procedures
2. Age: Female and/or male aged >18 years
3. Subject must have type 1 diabetes (as diagnosed clinically) ≥ 12 months
4. HbA1c <10 %
5. Insulin use with an average daily dose between 0.6 - 2.0 U/kg administered by insulin pump (CSII)
6. BMI 23.0 to 35.0 kg/m2 minimum weight of 50 kg
7. Women of childbearing potential (WOCBP) must be using an acceptable method of contraception to avoid pregnancy throughout the study as judged by the investigator
8. WOCBP must have a negative serum pregnancy test at screening as well as negative urine tests at follow up visits
9. Women must not be breastfeeding

Exclusion Criteria:

1. Target Disease Exclusions

   1. History of T2DM (type 2 diabetes mellitus), maturity onset diabetes of young (MODY), pancreatic surgery or chronic pancreatitis
   2. Any use of oral hypoglycemic agents within 2 weeks prior to the screening visit
   3. History of diabetes ketoacidosis (DKA) within 12 weeks prior to prior to the screening visit
   4. History of diabetes insipidus
   5. History of hospital admission for glycemic control (either hyperglycemia or hypoglycemia) within 3 months prior to prior to the screening visit
   6. Frequent episodes of hypoglycemia as defined by more than one episode requiring assistance, emergency care (paramedics or emergency room care) or glucagon therapy (in children defined as seizure or loss of consciousness) , or more than 2 unexplained episodes of symptomatic hypoglycemia within 3 months prior to the screening visit.

      An unexplained event is defined as an event that cannot be explained by circumstances such as dietary (e.g. missed meal), strenuous exercise, error in insulin dosing, etc.
   7. Hypoglycemic unawareness
   8. History of Addison's disease or chronic adrenal insufficiency
2. Physical and Laboratory Test Findings

   1. Random C-Peptide >0.5 nmol/l
   2. Aspartate aminotransferase (AST) > 2X Upper limit of normal (ULN)
   3. Alanine aminotransferase (ALT) > 2X ULN
   4. Serum total bilirubin > 2X ULN (except known Gilbert's disease)
   5. Creatine kinase (CK) > 3X ULN
   6. Estimated GFR (eGFR) by the Modification of Diet in Renal Disease (MDRD) formula ≤ 60 ml/min/1.73m2. The renal function, eGFR will be estimated by the abbreviated MDRD, using laboratory measurements of serum creatinine collected at screening
   7. Hemoglobin ≤ 11.0 g/dl (110 g/l) for men; hemoglobin ≤10.0 g/dl (100 g/L) for women.
   8. Positive for hepatitis B surface antigen or anti-hepatitis C virus antibody or HIV in patient's history.
   9. Abnormal Free T4 Note: abnormal TSH value at screening will be further evaluated for free T4.Subjects with abnormal free T4 values will be excluded. A one-time retest may be allowed, as determined by the Investigator, after a minimum of 6 weeks following the adjustment of thyroid hormone replacement therapy in subject who have had a prior diagnosis of a thyroid disorder and who are currently receiving thyroid replacement therapy. Such cases should be discussed with the Sponsor prior to re-testing. The subject must have all screening procedures and laboratory assessments performed as part of this re-test, and all of these must meet enrolment eligibility criteria. The subject's number will, however, remain the same as initially assigned.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-08-26 (Actual)

PRIMARY OUTCOMES:
time to development of DKA | 12 hours
  time from Insulin withdrawal to development of DKA (defined as HCO3 -< 19mmol/L)

SECONDARY OUTCOMES:
time to decrease of ph level | 12 hours
  time from Insulin withdrawal to decrease of pH < 7.30

CONTACTS AND LOCATIONS:
Overall Officials: Torben Biester, MD, Principal Investigator — Kinderkrankenhaus auf der Bult
Locations (1):
- Kinder- und Jugendkrankenhaus AUF DER BULT, Hanover, Lower Saxony, Germany